CLINICAL TRIAL: NCT00394498
Title: Stem Cell Mobilization by G-CSF by Granulocyte Colony Stimulating Factor Post Myocardial Infarction to Promote Myocyte Repair
Brief Title: Stem Cell Mobilization by G-CSF Post Myocardial Infarction to Promote Myocyte Repair
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 135287
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Stem Cells
MeSH Terms: conditions — Myocardial Infarction | interventions — Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor

SUMMARY:
Eighty-six patients with heart attacks will be identified at our hospital. Post heart attack we will assess heart function, blood flow to the heart, and heart cell function. We will assess these parameters using nuclear cardiology scans that are used in everyday cardiology practice. The patients will then be divided into 2 groups. One group will receive a medication called G-CSF and the other group will receive a placebo. We will give this drug (1-2ml) for 4 days beneath the skin. We will take the patients blood during this time and measure how the drug affected their blood. The patients will all have the nuclear cardiology tests again in 6 weeks and 6 months to see how their heart is functioning. As well, they will have a six month angiogram. All the patients will otherwise receive optimal care from their Cardiologist. They will be seen at 6, 12, 24, and 52 weeks to assess them clinically.

This study will test the effects of G-CSF on the heart function of patients who have had a heart attack. It is a medication that that has been shown in an animal model to improve heart function after a heart attack. It is a medication that has been used for many years to treat patients with cancers and to increase the number of cells donated by healthy bone marrow donors. It has no serious side effects. It works by increasing the number of a person's own stem cells in the blood. Stem cells are special cells that are present in our bodies that have the ability to form new cells. It had been thought that the heart could not make new cells after it has been damaged. Other investigators have shown that this might not be the case. It is now thought that after an injury, stem cells from the bone marrow can transform into cells of the injured tissue. Therefore, we are trying to increase the number of stem cells in the circulation with G-CSF so as to increase repair in the heart after it has been damaged. This strategy has never been tried in human beings and if successful could greatly reduce death and suffering from heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Large anterior wall ST elevation AMI defined by: Post AMI LVEF less than 45% as assessed by echocardiography. It is standard practice at our institution to obtain echocardiograms on such patients before day 4 post AMI.
2. Age between 40 -75 years
3. Angiographically patent infarct related artery (IRA) with TIMI 3 flow with no significant stenosis (>70% diameter stenosis in non-intervened upon arteries or >30% in arteries that had PTCA), no dissection or visible thrombus, and considered at low risk for re-occlusion by the Cardiologist performing the coronary angiography. In patients who have undergone PTCA, this assessment will be none on a post PTCA angiogram. This will be the majority of patients.
4. Eligible for treatment with G-CSF within the 5 days Post AMI.

Exclusion Criteria:

1. Prior STEMI
2. Patients with regional wall motion abnormalities in the non-infarct region
3. Prior CABG or need for CABG
4. Patients with significant valve disease; defined as stenosis or regurgitation graded as greater than moderate (2+).
5. Patients with clinically apparent, concurrent infection, requiring intravenous antibiotics
6. Patients who are or could be pregnant
7. Patients with another etiology of LV dysfunction (known/suspected non ischemic cardiomyopathy, previous anthracycline therapy, known ethanol abuse (greater than 6 oz. ethanol/day on a regular basis).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2005-09; Study Completion 2006-10

PRIMARY OUTCOMES:
6 month Left ventricular ejection fraction

SECONDARY OUTCOMES:
6 week left ventricular ejection fraction
6 week myocardial FDG-PET uptake
6 week myocardial Ammonia-PET perfusion
6 week/month left ventricular diastolic volume
6 week/month left ventricular systolic volume

CONTACTS AND LOCATIONS:
Overall Officials: Chris A Glover, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Hibbert B, Hayley B, Beanlands RS, Le May M, Davies R, So D, Marquis JF, Labinaz M, Froeschl M, O'Brien ER, Burwash IG, Wells GA, Pourdjabbar A, Simard T, Atkins H, Glover C. Granulocyte colony-stimulating factor therapy for stem cell mobilization following anterior wall myocardial infarction: the CAPITAL STEM MI randomized trial. CMAJ. 2014 Aug 5;186(11):E427-34. doi: 10.1503/cmaj.140133. Epub 2014 Jun 16. PMID 24934893
- [Derived] Anselm DD, Anselm AH, Renaud J, Atkins HL, de Kemp R, Burwash IG, Williams KA, Guo A, Kelly C, Dasilva J, Beanlands RS, Glover CA. Altered myocardial glucose utilization and the reverse mismatch pattern on rubidium-82 perfusion/F-18-FDG PET during the sub-acute phase following reperfusion of acute anterior myocardial infarction. J Nucl Cardiol. 2011 Aug;18(4):657-67. doi: 10.1007/s12350-011-9389-5. Epub 2011 May 13. PMID 21567283